CLINICAL TRIAL: NCT04758702
Title: The Clinical Impact of L-PRF, H-PRF or the Use of Surgical Stent on Palatal Donor Site Healing: A Randomized, Three Parallel Arms Clinical Trial.
Brief Title: The Clinical Impact of L-PRF, H-PRF or the Use of Surgical Stent on Palatal Donor Site Healing.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abdo Y Ismail (Other)
Responsible Party: Sponsor-Investigator, Abdo Y Ismail, Post-graduate Periodontics Resident, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 63364
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Lack of Keratinized Gingiva

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP 1 (Experimental): L-PRF membranes will be placed on the palatal donor site to help stabilizing the blood clot and release of growth factors that help in deceasing the discomfort wound healing.
  Interventions: Biological: L-PRF (Leucocyte- platelet rich fibrin)
- GROUP 2 (Experimental): H-PRF membranes will be placed on the palatal donor site to help stabilizing the blood clot and release of growth factors that help in deceasing the discomfort wound healing.
  Interventions: Biological: H-PRF (Horizontal -platelet rich fibrin)
- GROUP 3 (Experimental): A surgical stent will be delivered to cover the surgical site and apply pressure on the wound site.
  Interventions: Device: Surgical stent

INTERVENTIONS:
Biological: L-PRF (Leucocyte- platelet rich fibrin) — Leucocyte-Platelet rich fibrin is a high density fibrin clot. it serves as a biological healing matrix by supporting cell migration and cytokine release, expanding the range of its potential applications greatly. Patient's own blood is centrifuged using (Intra-spin) FDA approved centrifuge on 45 degrees angle on 2700 rpm for 12 minutes.
  Arms: GROUP 1
Biological: H-PRF (Horizontal -platelet rich fibrin) — Platelet rich fibrin is a high density fibrin clot. it serves as a biological healing matrix by supporting cell migration and cytokine release, expanding the range of its potential applications greatly.Horizontally centrifuged platelet rich fibrin using (Bio-prf) centrifuge on 700 g force for 8 minutes. On a horizontal centrifugation, the cells separate much more efficiently throughout the entire membrane. This leads to better layer separation and also favors cells that are evenly distributed throughout the PRF clot.
  Arms: GROUP 2
Device: Surgical stent — An essix surgical stent will be obtained using a high vacuum suction and used to protect the denuded donor site after suturing the wound. (Biostar® Scan/Biostar®V) will be used to make the stent.
  Other Names: Essix retainer
  Arms: GROUP 3

SUMMARY:
A Randomized, Three Parallel Arms Clinical Trial to evaluate s the clinical impact of L-PRF vs H-PRF vs Palatal stent on the healing of the donor palatal site.

DETAILED DESCRIPTION:
A Randomized, Three Parallel Arms Clinical Trial. The primary objective is to assess the clinical impact of L-PRF vs H-PRF vs Palatal stent on the healing of the donor palatal site by comparing the percentage of re-epithelization of the palatal donor site at 5, 10, 14 and 21 days using a standardized intraoral palatal photo.

The secondary objective is to compare the post op discomfort between the three groups during the healing period daily for 2 weeks using the Visual Analogue Scale (VAS) and Analgesic consumption.

All subjects from the University of Kentucky College of Dentistry clinics. Subjects that are coming increasing the width of keratinized tissue or for the treatment of gingival recession, and match the inclusion criteria will be told about the research and offered the opportunity to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 18-65 years of age.
2. Subjects need FGG or de-epithelialized Connective tissue graft
3. Good oral hygiene (Plaque and bleeding indexes <20%).
4. Subjects can withstand alginate impression or wear a retainer.
5. No other surgery or need for analgesics at the same site.

Exclusion Criteria:

1. Subjects with any systemic disorders that might compromise wound healing (Uncontrolled diabetes mellitus, rheumatoid arthritis, osteoporosis, chemotherapy/radiotherapy and immunological disorders).
2. Smokers
3. Patients not maintaining oral hygiene (plaque score >20%)
4. Pregnant or breastfeeding females.
5. Inability to provide informed consent.
6. Grafts thickness more than 2mm will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
The Clinical Impact of L-PRF, H-PRF, or the Use of a Surgical Stent on Palatal Donor Site Healing. | 5 days
  The primary outcome is to asses the percentage of re-epithelization of the palatal donor site and assess primary wound healing.
The Clinical Impact of L-PRF, H-PRF, or the Use of a Surgical Stent on Palatal Donor Site Healing. | 10 days
  The primary outcome is to asses the percentage of re-epithelization of the palatal donor site and assess primary wound healing.
The Clinical Impact of L-PRF, H-PRF, or the Use of a Surgical Stent on Palatal Donor Site Healing. | 14 days
  The primary outcome is to asses the percentage of re-epithelization of the palatal donor site and assess primary wound healing.
The Clinical Impact of L-PRF, H-PRF, or the Use of a Surgical Stent on Palatal Donor Site Healing. | 21 days
  The primary outcome is to asses the percentage of re-epithelization of the palatal donor site and assess primary wound healing.

SECONDARY OUTCOMES:
The Clinical Impact of L-PRF, H-PRF, or the Use of a Surgical Stent on Palatal Donor Site Healing. | 5 days
  The secondary outcome is to compare the post-operative discomfort between the three groups during the healing period using the Visual Analogue Scale and Analgesic consumption. The visual analog scale is a validated, subjective measure for acute and chronic pain; with (0) indicates no pain and (10) indicates worst pain possible. Scores will be recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain", which is the (0) and "worst pain possible", which is the (10). Also, the patient will write down his/her analgesic consumption, including the frequency and the amount used.
The Clinical Impact of L-PRF, H-PRF, or the Use of a Surgical Stent on Palatal Donor Site Healing. | 10 days
  The secondary outcome is to compare the post-operative discomfort between the three groups during the healing period using the Visual Analogue Scale and Analgesic consumption. The visual analog scale is a validated, subjective measure for acute and chronic pain; with (0) indicates no pain and (10) indicates worst pain possible. Scores will be recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain", which is the (0) and "worst pain possible", which is the (10). Also, the patient will write down his/her analgesic consumption, including the frequency and the amount used.
The Clinical Impact of L-PRF, H-PRF, or the Use of a Surgical Stent on Palatal Donor Site Healing. | 14 days
  The secondary outcome is to compare the post-operative discomfort between the three groups during the healing period using the Visual Analogue Scale and Analgesic consumption. The visual analog scale is a validated, subjective measure for acute and chronic pain; with (0) indicates no pain and (10) indicates worst pain possible. Scores will be recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain", which is the (0) and "worst pain possible", which is the (10). Also, the patient will write down his/her analgesic consumption, including the frequency and the amount used.
The Clinical Impact of L-PRF, H-PRF, or the Use of a Surgical Stent on Palatal Donor Site Healing. | 21 days
  The secondary outcome is to compare the post-operative discomfort between the three groups during the healing period using the Visual Analogue Scale and Analgesic consumption. The visual analog scale is a validated, subjective measure for acute and chronic pain; with (0) indicates no pain and (10) indicates worst pain possible. Scores will be recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain", which is the (0) and "worst pain possible", which is the (10). Also, the patient will write down his/her analgesic consumption, including the frequency and the amount used.

CONTACTS AND LOCATIONS:
Overall Officials: Mohanad Al-Sabbagh, DDS, MS, Study Chair — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No